CLINICAL TRIAL: NCT06019390
Title: eHealth for Screening Health Risks in Home-Based Older Adults: A Prospective Observational Study
Brief Title: eHealth for Screening Health Risks in Home-Based Older Adults: A Prospective Study
Acronym: Proxi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Presage (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Presage_Proxi
Record Dates: First submitted 2023-08-21; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Frail Elderly Syndrome; Older
Keywords: screening tool; prevention; artificial intelligence; geriatric syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental)
  Interventions: Device: Presage care

INTERVENTIONS:
Device: Presage care — A screening questionnaire completed by the family caregiver focused on functional and clinical autonomy of the patient (ie, activities of daily life), possible medical symptoms (eg, fatigue, falls, and pain), changes in behavior (eg, recognition and aggressiveness), and communication with relative or their surroundings.

SUMMARY:
Introduction: Due to the worldwide ageing population and the increasing prevalence of chronic illnesses and cognitive deficits, appropriate instruments for frailty early screening and assessment of geriatric syndromes are required. Digital tools based on artificial intelligence can help improve the evaluation and screening of health risks in the older adults.

Objectives: This study aims to evaluate the effectiveness of the PRESAGE CARE questionnaire in screening geriatric syndromes among older adults and to assess its correlation with standardized test scores of the comprehensive geriatric assessment (CGA).

Methods: A monocentric prospective observational study will be conducted between October 2023 and July 2024, on seniors who are in the day hospitalization service of Charles-Foix hospital in France. During the consultation with older adults, the investigators will ask the patient's home caregiver to use the PRESAGE CARE application to fill in the PRESAGE CARE questionnaire. Once the questionnaire will be completed on the application, the PRESAGE platform will automatically recorde specific risks for each senior. Subsequently, the investigators will retrieve the data from standardized tests conduct on the same day and enter the results for each patient into the platform.

The primary outcome will be the correlation between standardized test scores and the risks computed by the Presage Care system for the risk of depression, the risk of undernutrition, the risk of cognitive impairment and the risk of loss of autonomy in activities of daily living.

Secondary outcome will be the comparison of the Area Under the Median Curve (AUC), and the sensitivity, specificity and positive predictive values of artificial intelligence (AI)-based models on the Présage Care questionnaire.

DETAILED DESCRIPTION:
During the consultation and the assessment of the older adult by the physicians and the nurses at the day hospitalization service of the hospital, patient's relative fill out PRESAGE CARE questionnaire. Then, the investigators retrieved the data from the standardized tests completed the same day by the health professionals and filled in the test results for each patient on the platform.

ELIGIBILITY:
* Inclusion criteria :

  1. family members of individuals aged 65 and above,
  2. who are present within the day hospitalization service of Charles-Foix Hospital
  3. and able to provide informed consent.
* Non inclusion criteria

  1. refuse to give their consent to participate in the study,
  2. or have cognitive impairments
  3. or are occasional caregivers.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlationbetween standardized test scores and the corresponding risks identified by PRESAGE questionnaire. | 6 months
  Kendall's correlation coefficient (Tau test) will be used to analyze the correlation between the risks calculated by the Présage Care algorithm and the results of the associated standardized scale.

SECONDARY OUTCOMES:
predictive performance of Presage Care questionnaire for health risk detection | 6 months
  For secondary outcoumes, the Chi2 test will be used to compare the high-risk rate and the diagnostic rate for each risk. Presage Care risks will be represented as binary Yes/No variables (at risk/no risk) or as ordinal variables (different levels of risk). Scores on the standardized MNA, GDS15 and MMSE tests will be grouped into binary variables according to the threshold for each test described in the literature, with 0 = "normal" score. For the IADL and ADL scales, the threshold defined represents total autonomy (independence in each of the domains scored). Predictive performance will be assessed by the median area under the curve, sensitivity, specificity, positive predictive value, negative predictive value, Youden index, for each Presage risk with the associated scale score. Data analysis will be performed using R studio (version 2022.07.2+576) and Python software.

IPD SHARING:
Plan to Share IPD: No